CLINICAL TRIAL: NCT02513225
Title: Randomized Controlled Trial of an Adapted STD Screening and Risk Reduction Intervention
Brief Title: Trial of an Adapted STD Screening and Risk Reduction Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14020838
Record Dates: First submitted 2015-07-09; First posted 2015-07-31 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Use; Drug Use; Diagnostic Self Evaluation; Gonorrhea; Unprotected Sex; Chlamydia; Trichomonas
MeSH Terms: conditions — Alcohol Drinking; Gonorrhea; Unsafe Sex; Chlamydia Infections; Trichomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The adapted Project EMPWR will be comprised of 2 sessions delivered approximately 7-10 days apart by a trained Apache paraprofessional interventionist. In the first session, interventionists will use curriculum to help participants understand their personal risk factors for STDs including HIV/AIDS (i.e., substance use, mental and emotional health, sexual health, etc.) and develop an achievable personalized risk-reduction plan that emphasizes individual and community-based strengths and resources.The second counseling session will consist of the disclosure of results (if tested) and the provision of social support to help participants develop a longer-term risk-reduction plan. At visit two, participants in both groups will be offered a STD screening protocol test.
  Interventions: Behavioral: Project EMPWR; Other: Optimized Standard Care (OSC)
- Control (Other): The comparison condition will consist of Optimized Standard Care (OSC) alone. All participants will receive OSC at the first visit. OSC includes the distribution of educational pamphlets and provision of information on substance use, signs and symptoms of mental health problems, and information about STD screening resources. At visit two, participants in both groups will be offered a STD screening protocol test.
  Interventions: Other: Optimized Standard Care (OSC)

INTERVENTIONS:
Behavioral: Project EMPWR — Participants will receive both Adapted Project EMPWR and Optimized Standard Care (OSC).
  Other Names: Intervention Condition
  Arms: Intervention
Other: Optimized Standard Care (OSC) — Participants will receive Optimized Standard Care (OSC) alone.

SUMMARY:
The goal of this research study is to evaluate the impact of a paraprofessional-delivered, culturally adapted, evidence-based intervention (EBI) on sexually transmitted disease (STD), substance use and poor mental/emotional health among American Indians (AI) through a Randomized Controlled Trial (RCT). These intertwining risks have produced marked disparities and have unique cultural and social determinants in Native communities. If aims are achieved, scientific knowledge and community-based practice will be advanced in areas vital to AI communities, and to STD and drug prevention science.

Prior to this study, the investigators applied findings from research protocol (IRB#00005929) and adapted a brief intervention to reduce risk and increase protective behaviors for STDs, HIV/AIDS, substance use and poor mental/emotional health, and to promote STD screening. The specific aim of the current study is to compare the efficacy of the adapted brief intervention vs. a comparison condition on participants' condom use, STD screening and treatment-seeking behaviors, substance use and emotional/mental health outcomes at 3 and 6 months post-intervention.

DETAILED DESCRIPTION:
STDs including Neisseria gonorrhea, Chlamydia trachomatis and Trichomonas vaginalis, are an urgent problem in American Indian/Alaska Native (AI/AN) communities due to a constellation of risk and contextual factors affecting tribal populations. Geographic isolation and cultural and social stigmatization contribute to poor access to screening, counseling and education, and diminished opportunities for early identification of STDs. Evidence-based prevention, STD screening and early identification are the best public health strategies to address a potential epidemic among AI/ANs. However, there is currently a paucity of such strategies that have been demonstrated in AI/AN populations. An intervention targeting STD screening and related risk reduction behaviors has the potential to circumvent the continuous transference of disease.

Participating Community: The Fort Apache Reservation is home to ~17,000 White Mountain Apache tribal members, with almost half <20 years of age. The reservation encompasses 1.7 million acres along northeastern Arizona. The Tribe endures notable demographic and environmental challenges that impact behavioral risks among community members: 61% of the population >16 years old are either "Not in Labor Force" or unemployed. 47% of Apaches aged ≥25 have not received a high school diploma. The median household income is $26,973 and 47% of the population lives below the federal poverty line. Over half (53%)(1) of all Apache households are led by single mothers;(2) 75% of children are born to unwed mothers.(3) These factors contribute to high rates of school drop-out, substance use, high-risk sexual behavior and poor mental and emotional health in the void of effective interventions. Despite these challenges, the Apache community has successfully demonstrated the ability to adapt and implement effective paraprofessional-administered interventions.(4,5)

Epidemiology of STD and Related Risk Behaviors: Recently, STD rates have increased throughout Arizona, and the state's AI population bears a disproportionately high burden of new infections.(6) In 2011, the chlamydia rate among AIs in Arizona was 6 times the rate for non-Hispanic Whites.(6) The rate of gonorrhea among AIs in Arizona tripled between 2009 and 2011, a rise largely attributed to "outbreaks in tribal areas in the northeastern quadrant of Arizona."(6) In 2011-2012, the chlamydia rate among Apaches was 2,116/100,000 for all ages, nearly 5 times both Arizona and national all-ages rates. The Apache gonorrhea rate was 749/100,000 for all ages in 2011-2012, approximately 7 and 10 times higher than national and Arizona all-ages rates, respectively. Previous studies indicate that among all races and ethnicities AI/ANs have some of the highest rates of inconsistent condom use, multiple sex partners and early sexual initiation.(7-10) The intersection of several behavioral risks such as poor mental health, drug use and binge alcohol use has shown to increase STD risk behaviors. A study conducted with Apache teens with recent suicidal behavior revealed high rates of lifetime drug use: 92% for alcohol, 88% for marijuana, 38% for crack/cocaine, and 35% for methamphetamines, which is 3 times that of all AI/AN adolescents in 2009. Highlighting the intersection of risk, 48% of those that were sexually active had ever used cocaine compared with 17% of those not sexually active; similarly, 40% of sexually active participants had ever used methamphetamine compared with 17% of participants that were not sexually active.

There have been scarce rigorous RCTs of behavioral health interventions among AI populations and none that have analyzed an EBI promoting STD screening or addressing the interrelated risks of substance use, poor emotional health and STDs/ HIV/AIDS. This study targets the shared root causes of substance use and sexual risk behaviors and aims to develop personalized, strengths-based risk reduction strategies tailored to participants' and the community's specific risk profiles.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified adults of American Indian ethnicity, who are members of the White Mountain Apache community
* Ages 18 to 49;
* Written informed consent to participate in the study;
* Currently sexually active;
* At least one episode of binge substance use or suicidal ideation recorded in the Apache community-based surveillance system in the past 90 days;
* Participant must agree to be audio recorded during intervention sessions

Exclusion Criteria:

* Inability to participate in full intervention (e.g., planned move, residential treatment, etc.)
* Severe risk for suicide (i.e., suicide attempt within past 6 months) or
* Unwilling to be randomized

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Self reported condom use | 6 months
  Change in self reported condom use at last sex, between intervention and control groups between baseline and 6 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Tingey, MPH/MSW, Principal Investigator — Center for American Indian Health
Locations (1):
- Fort Apache Reservation, Fort Apache, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chambers R, Tingey L, Beach A, Barlow A, Rompalo A. Testing the efficacy of a brief sexual risk reduction intervention among high-risk American Indian adults: study protocol for a randomized controlled trial. BMC Public Health. 2016 Apr 29;16:366. doi: 10.1186/s12889-016-3040-y. PMID 27129956